CLINICAL TRIAL: NCT03653169
Title: Use of Transcranial Magnetic Stimulation to Reduce Craving for Individuals With Opioid Use Disorder Taking Buprenorphine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Heather Burrell Ward, Resident Physician in Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100313439
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Opioid-use Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Open-Label Active TMS (Experimental): All subjects will receive open-label treatment with active Transcranial Magnetic Stimulation (TMS)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — TMS is a form of noninvasive brain stimulation. An external electromagnetic coil is placed on the head, and a large current is passed through an insulated wire coil held flat on the surface of a subject's scalp in a fraction of a millisecond. This pulse of current induces a weak electrical current within the surface brain cortex. Repetitive trains of TMS pulses (repetitive TMS or rTMS) can transiently modulate corticospinal excitability following the rTMS train. When current is delivered at high frequency (10 Hz), it may simultaneously increase the activity of the brain at this site. In this study, individuals will receive 10 treatments with intermittent theta burst stimulation (twice daily for 5 days).

SUMMARY:
The aim of this study is to investigate the effects of transcranial magnetic stimulation (TMS) on craving in individuals treated with buprenorphine for opioid use disorder. In this study, individuals will receive 10 sessions of TMS (twice daily for 5 days). The investigators will assess craving, substance use, and mood throughout the study and 1-2 weeks post-treatment.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of transcranial magnetic stimulation (TMS) on craving in individuals treated with buprenorphine for opioid use disorder. Investigators will enroll subjects aged 18-65 years old who are currently in treatment with buprenorphine for opioid use disorder. Included subjects will have initiated treatment with buprenorphine in the last 3 months, be able to read, write, and understand English, and, if female, agree to use contraception. Subjects will be excluded if they have a history of bipolar or psychotic illness, current depression, use substances other than opioids, take medications that lower seizure threshold or impair neuroplasticity, have chronic pain, have a history of seizure or any other uncontrolled medical issue, or have a device or ferromagnetic implant in the head or neck. Enrolled subjects will receive 10 (twice daily for 5 days) sessions of active TMS (intermittent theta burst stimulation) to the left dorsolateral prefrontal cortex (L DLPFC) on consecutive weekdays. Investigators will assess craving, substance use, and mood throughout the study and 1-2 weeks post-treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old
* Initiated treatment with buprenorphine for opioid use disorder within the last 3 months
* Be able to understand, read and write English.
* If female and of childbearing age, agree to use acceptable birth control during the study treatment period (oral contraceptives, history of tubal ligation, history of a hysterectomy, or a reliable barrier method) during the study treatment period.

Exclusion Criteria:

* Lifetime history of bipolar disorder or psychotic disorder,
* Current depression as rated by PHQ-9 ≥ 20 (Kroenke, Spitzer, and Williams 2001, Suzuki et al. 2015)
* Moderate chronic pain (pain intensity rated ≥ 40 on 100-point VAS lasting at least 6 months (Stein et al. 2015)
* History of alcohol use disorder as rated by AUDIT-C ≥ 4 (at risk) (Babor et al. 2001)
* History of complicated withdrawal from alcohol (i.e. delirium tremens, seizure)
* Substance use disorder in the past year (other than opioid or nicotine), as assessed by drug screens,
* Neurologic disease including stroke, seizure, migraine, or severe head injury
* Major medical conditions that are not well-controlled or under the care of a physician
* Device (i.e. pacemaker, cochlear prosthesis, neurostimulator, intraocular metallic fragments) or ferromagnetic implant above the neck (within 30 cm of coil),
* Medication that lowers seizure threshold (i.e. immediate release bupropion, psychostimulants, tricyclic antidepressants) or impairs neuroplasticity (i.e. benzodiazepines)
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Cue-Induced Craving, as measured by 0-100 Visual Analog Scale | End of TMS Treatments (1 week)
  Visual Analog Scale (0-100, where 0 = no craving, 100 = maximum craving)
Drug Craving, as measured by 0-100 Visual Analog Scale | End of TMS Treatments (1 week)
  Visual Analog Scale (0-100, where 0 = no craving, 100 = maximum craving)

SECONDARY OUTCOMES:
Opioid Use and Relapse, as measured by Timeline Followback Calendar (days of opioid use) | End of TMS Treatments (1 week)
  Timeline Followback calendar, which measures days of opioid use over the past 2 weeks
Retention in Buprenorphine Treatment | End of TMS Treatments (1 week)
  Treatment Retention: subjects actively engaged in buprenorphine treatment, attending appointments
Symptoms of Depression, as measured by the Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) | End of TMS Treatments (1 week)
  Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16), where higher score indicates more severe depressive symptoms
Drug Craving, as measured by 0-100 Visual Analog Scale | 1-2 weeks after completion of TMS treatments
  Visual Analog Scale (0-100, where 0 = no craving, 100 = maximum craving)
Opioid Use and Relapse, as measured by Timeline Followback Calendar (days of opioid use) | 1-2 weeks after completion of TMS treatments
  Timeline Followback calendar, which measures days of opioid use over the past month
Retention in Buprenorphine Treatment | 1-2 weeks after completion of TMS treatments
  Treatment Retention: subjects actively engaged in buprenorphine treatment, attending appointments
Symptoms of Depression, as measured by the Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) | 1-2 weeks after completion of TMS treatments
  Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16), where higher score indicates more severe depressive symptoms
Neuropsychologic Testing Battery | End of TMS treatment (1 week)
  Penn Computerized Neuropsychologic Battery
Impulsivity | End of TMS treatment (1 week)
  Barratt Impulsivity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Ward, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No